CLINICAL TRIAL: NCT00983359
Title: A Phase II Trial of Focal Therapy in the Treatment of Patients With 1-3 Brain Metastases
Brief Title: Stereotactic Radiation Therapy in Treating Patients With Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Mario Ammirati, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-06138; NCI-2011-03139 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: tumors metastatic to brain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (conformal stereotactic radiation therapy) (Experimental): Patients undergo conformal stereotatic radiation
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Patients undergo conformal stereotatic radiation therapy QD (every day) over 5 days.
  Other Names: Radiation

SUMMARY:
RATIONALE: Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This phase II trial is study how well stereotactic radiation therapy works in treating patients with brain metastases

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the neurological death rate following the initiation of conformal stereotactic radiotherapy in patients with 1-3 brain metastases.

Secondary

* To determine the overall survival rate at 6 months.
* To determine the progression-free survival rate or brain metastases recurrence rate at 6 months.
* To determine the time to neurological death, time to systemic death, and Karnofsky decay time.
* To determine the frequency and severity of adverse events associated with conformal stereotactic radiotherapy.

OUTLINE: Patients undergo conformal stereotactic radiotherapy over 5 days to an area including 3 mm around the metastases or the surgical cavity. Patients may receive additional radiotherapy if symptomatic metastases emerge at different sites.

After completion of study treatment, patients are followed up at 1 and 2 months and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histology-confirmed cancer with 1 to 3 symptomatic brain metastases imaged by MRI/CT scans.
* Have cancer not originating in central nervous system (CNS)
* Karnofsky score of at least 60
* Given written consent
* At least 18 years of age

Exclusion Criteria:

* Prior whole brain radiotherapy or prior focal radiotherapy of the metastasis/es considered for this trial.
* Certain radiosensitive primary tumors such as small cell lung cancer, germ cell tumors, lymphoma, leukemia or multiple myeloma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Ammirati, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Ammirati M, Kshettry VR, Lamki T, Wei L, Grecula JC. A prospective phase II trial of fractionated stereotactic intensity modulated radiotherapy with or without surgery in the treatment of patients with 1 to 3 newly diagnosed symptomatic brain metastases. Neurosurgery. 2014 Jun;74(6):586-94; discussion 594. doi: 10.1227/NEU.0000000000000325. PMID 24589560
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment period was June 2007 to March 2010
Period: Overall Study
Arm/Group | Treatment (Conformal Stereotactic Radiation Therapy)
Started | 40
Not Eligible for Analysis | 1
Completed | 39
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Conformal Stereotactic Radiation Therapy)
Number analyzed (Participants) | 39
Age, Customized [Number; unit: patients]
  ≤60 | 20
  >60 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: patients]
  United States | 39
Extracranial metastases [Number; unit: patients]
  Absent | 19
  Present | 20
Number of brain metastases [Number; unit: patients with brain metastases] — Patients with ≥4 brain metastases were eligible for study if only 1 to 3 were symptomatic and all others asymptomatic.
  patients with brain metastases
    1 | 25
    2 | 4
    3 | 8
    ≥4 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Dying of Neurological Death, Defined as Dying With Progressive Neurological Dysfunction Regardless of Systemic Disease Status
Description: Neurological death is defined as dying with progressive neurological dysfunction regardless of systemic disease status. Patients wtih severe neurological disability who die of intercurrent illness will also be considered to have died of neurological death.
Time Frame: Up to 5 years
Measure: Number; unit: patients
Arm/Group | Treatment (Conformal Stereotactic Radiation Therapy)
Number analyzed (Participants) | 39
patients | 5

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from enrollment to first date of progressive or recurrent disease. Worsening of neurological symptoms is considered indicative of neurological disease progression. Patients who die of disease-related or treatment-related causes will be considered to have progressed at their date of death; i.e., not be considered 'censored'. PFS will be considered censored only if no progression is noted or if the patient dies of a clearly non-cancer-related event such as accident.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Conformal Stereotactic Radiation Therapy)
Number analyzed (Participants) | 39
months | 11 [4 to 21]

3. Secondary Outcome: Time to Neurological Death
Description: Time from enrollment to date of death directly due to brain metastases. Deaths from other causes including hemorrhage or infection will be considered 'censored' observations in the setting of neurologic improvement or stabilization. If the patient dies of any cause with worsening of neurologic symptoms, the death will be counted as an 'event' or neurological death.
Time Frame: From time of enrollment up to 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Conformal Stereotactic Radiation Therapy)
Number analyzed (Participants) | 5
months | 13 [5 to 18]

4. Secondary Outcome: Time to Systemic Death
Description: Descriptive analysis will be conducted using Kaplan-Meier survival analysis
Time Frame: From time of enrollment up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Conformal Stereotactic Radiation Therapy)
Number analyzed (Participants) | 39
months | 16 [9 to 24]

5. Secondary Outcome: Karnofsky Decay Time
Description: Time from enrollment to the date the patient's Karnofsky performance score drops below 60. If the patient dies of any cause with no documentation of a drop in their Karnofsky score to less than 60, the date of death will be used as the date of worsening of the Karnofsky score. A patient with a Karnofsky score of 60 or greater requires occasional assistance, but is able to care for most of his/her needs. A patient's Karnofsky decay time will be considered censored if the patient is still under follow up with a Karnofsky score of 60 or greater and if the patient dies of a non-cancer-related cause.
Time Frame: From time of enrollment up to 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Conformal Stereotactic Radiation Therapy)
Number analyzed (Participants) | 39
months | 14 [1 to 62]

ADVERSE EVENTS:
Description: The NCI Common Terminology Criteria for Adverse Events version 3 [CTCAEv3] was used to access adverse events for patients.
Arm/Group | Treatment (Conformal Stereotactic Radiation Therapy)
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes